CLINICAL TRIAL: NCT06084091
Title: Spectroscopic Assessment of Intramyocardial Oxygen Saturation During Open-Heart Surgery
Acronym: ECS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spectrocor (Industry)
Responsible Party: Sponsor
Other Study IDs: Safe-op 1.0 ECS
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Heart Valve Diseases
Keywords: monitoring, intraoperative; Heart Surgery
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Myocardial spectrometric measurement — Myocardial spectrometric measurement during open-heart Surgery

SUMMARY:
The goal of this observational study is to test in the safety and performance of intraoperative myocardial spectroscopic measurement in open-heart surgery patients

The main questions it aims to answer are:

* The Devices can record myocardial spectrometric data for analysis, and
* How these measures correlate with the occurring events, procedures, and clinical parameters during the operation.
* Number of participants with device-related adverse events as assessed by CTCAE v4.0

DETAILED DESCRIPTION:
The study design is based on measuring the depth of ischemia during the operation, which is compared to the intraoperative and postoperative morbidity of the patient, especially to the dysfunction of the heart. A qualified and experienced Monitor is assigned for the study to oversee and document the progress of the trial. The Monitor ensures the trial performance in accordance with the Protocol and Good Clinical Practice (GCP). The trial team conforms to ISO 13485 quality standards and ISO 14155 GCP. Processes included in the monitoring activities are documented in the quality management system. Below are described the summaries of all these activities. Source data will be collected and transferred into the electronic CRFs by site staff, and the collected data quality and the conformity to the Good Clinical Practice will be assessed by monitoring. Based on a risk assessment performed, a Data Monitoring Committee shall not be established. Clinical Research Associate (CRA) is responsible for checking the accuracy and completeness of Case Report Form (CRF) entries, source documents, and other investigation-related records against each other. Other responsibilities of CRA, including detailed Source Data Verification (SDV), are documented by the clinical project manager (CPM) or head of clinical research (HCR)(both are sponsor's representatives). SDVs will be performed and documented during monitoring visits. Monitoring planning, reporting, and visits are pre-defined and documented with pre-made templates per the sponsor's quality management system. Monitoring visits will be performed to cover data from all study participants, and according to QMS and the Standard Operation Procedures. The monitoring shall ensure that all source documentation is precise and document control is exercised in all relevant documentation. The monitoring ensures, that the Adverse events are always reported and appropriate authorities or stakeholders are informed.

ELIGIBILITY:
Inclusion Criteria:

* Any 18 to 90-year-old patient scheduled for an open-heart operation
* The ability to understand the study's objective and the risks involved.
* Informed consent obtained, including the agreement to authorization to use the protected personal patient records according to privacy legislation.

Exclusion Criteria:

* Inability to obtain an informed consent form
* Patients included as vulnerable population according to Finnish Medical Research Act, including retarded, pregnant women, nursing mothers, prisoners, or forensic patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for open-heart operation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial spectrometric recording | During operation
  Can the device record myocardial spectrometric data during open-heart surgery
Measurement correlation | During operation
  How the measurements correlate with the occurring events, procedures, and clinical parameters during the operation.

SECONDARY OUTCOMES:
Adverse event assessment | From admission to discharge, up to 2 weeks
  Assessment of the adverse events of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Raivio, PhD, Principal Investigator — Chief of Department, Head and Lung Center, Hospital District of Helsinki and Uusimaa
Locations (1):
- Heart and Lung Center, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No